CLINICAL TRIAL: NCT05965700
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1b/2a Study of NVG-291 in Spinal Cord Injury Subjects (CONNECT)
Brief Title: NVG-291 in Spinal Cord Injury Subjects
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NervGen Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NVG-291-201
Record Dates: First submitted 2023-07-16; First posted 2023-07-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Chronic Spinal Cord Injury; Subacute Spinal Cord Injury
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NVG-291 for Injection (Experimental): Injected under the skin (subcutaneous).
  Interventions: Drug: NVG-291
- Placebo (Placebo Comparator): Injected under the skin (subcutaneous).
  Interventions: Drug: NVG-291

INTERVENTIONS:
Drug: NVG-291 — A once daily injection

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Phase 1b/2a Study of NVG-291 in Spinal Cord Injury Subjects

DETAILED DESCRIPTION:
To evaluate the effect of NVG-291 on descending connectivity in subjects with subacute and chronic SCI (20 subjects per Cohort and results will be analyzed separately) using objective electrophysiological measures, in addition to clinical assessments. To evaluate safety and tolerability of NVG-291 in a SCI population, as measured by clinical assessments (Physical Examination, Vital Signs, ECG, etc.) as well as clinical laboratory measures. NOTE: Enrollment of the chronic cohort has been completed; approximately 20 individuals will be enrolled in the subacute group. For more information about the trial please visit www.connectscistudy.com.

ELIGIBILITY:
Inclusion Criteria:

A subject must provide written informed consent in accordance with local regulations prior to initiation of any study-specific activities/procedures. A legally authorized representative (LAR) may be used to assist in signing the informed consent.

Cervical SCI resulting from acute physical trauma.

Males and females

Age 18 - 75 years, inclusive.

Cervical SCI, incomplete, with a neurological level of injury being at C7 or higher.

Had incomplete cervical SCI within the period from 1 year to 10 years inclusive (Chronic cohort 1) OR within 20 days to 90 days inclusive (Subacute cohort 2) at time of randomization.

Must be able to volitionally initiate at least one step on one leg (without body weight support). (Cohort 1 only)

Must have a Walking Index for Spinal Cord Injury II (WISCI II) score as follows:

1. For Chronic cohort 1: Less than or equal to Level 14.
2. For Subacute cohort 2: Less than or equal to Level 10.

GRASSP/hand grip strength Prehension Ability score

For Chronic cohort 1:

i. Must have a score of at least 2 on at least one of the Prehension Ability grasp patterns of the GRASSP assessment in at least one upper extremity. ii. Must have no more than one Prehension Ability grasp patterns score = 4 in the upper extremity satisfying criterion i

For Subacute cohort 2:

i. Must have some voluntary (nonzero) force measured by grip dynamometry in at least one upper extremity.

ii. Must have no more than one Prehension Ability grasp patterns score = 3 in at least one upper extremity.

iii. Must not have a Prehension Ability grasp patterns score = 4 in the upper extremity satisfying criterion.

Presence of Motor Evoked Potentials (MEPs):

1. In two specific target muscle groups (Cohort 1)
2. In one specific target muscle group (Cohort 2)

Must be fluent in English.

Subjects must be willing and able to comply with scheduled visits, all sample collections, and other trial procedures.

Exclusion Criteria:

Nontraumatic SCI (e.g., due to infection, ischemia, metabolic abnormality, congenital abnormality, malignancy, radiation injury, surgical complications, or other disease process).

Spinal cord injury due to gunshot wound or penetrating injury.

Two or more (noncontiguous) spinal cord lesions.

MRI or CT evidence of anatomically complete spinal cord transection.

Any form of ventilatory dependence.

Any condition that precludes adequate clinical assessment of all four extremities, such as contracture, peripheral nerve injury, amputation.

History of uncontrolled seizures or any seizure within the last 6 months (Cohort 1). History of uncontrolled seizures, or any seizure occurring 1 week or more after the SCI (Cohort 2)

Metal implant in the head that is likely to interfere with MRI analysis.

Pregnant or breast feeding.

Any neurological condition that is considered to interfere with performance or likly confound assessment, such as multiple sclerosis, stroke, or progressive syringomyelia.

History of substance abuse within 12 months prior to screening, based on medical records or self-report.

Evidence of spinal instability or persistent spinal stenosis and/or compression related to initial trauma.

Prior treatment with cell therapy delivered into the CNS (intrathecal or intraparenchymal).

Severe neuropathic pain inadequately controlled by medication.

Body mass index (BMI) > 40 (body weight in kilograms divided by height in meters squared).

Received botulinum toxin injection(s) in an upper or lower extremity muscle in the prior 6 months.

Received 4-aminopyridine within 7 days of first dose..

Prior treatment with a protein tyrosine phosphatase sigma (PTPσ) mimetic peptide.

Intrathecal opioid use.

Currently participating in an interventional clinical trial.

Received a non-permitted medication within 5.5 half-lives or 7 days, whichever is longer, prior to randomization

Receiving any treatment intended to enhance neuroplasticity (e.g., electrical stimulation, acute intermittent hypoxia) at the time of consent to participate in this study or within 4 weeks of randomization, whichever is longer.

Any implanted internal spinal cord stimulator.

Currently receiving neuromuscular stimulation.

Currently receiving vagal or phrenic nerve stimulation.

Chronic cohort 1 only: Any contraindication to undergo baseline and on study MRIs such as:

1. History of a cardiac pacemaker or pacemaker wires, OR
2. Ferromagnetic metallic particles in the body, OR
3. Baclofen pump, OR
4. Vascular clips in the head, OR
5. Prosthetic heart valves, OR
6. Severe claustrophobia impeding ability to participate in an imaging study.

Malignancy within 5 years prior to screening, except for non-melanoma skin cancers or cervical or breast ductal carcinoma in situ.

History of medically significant hepatic disease or evidence of impaired liver function based on initial laboratory testing

Severe renal insufficiency, as defined by eGFR < 30 mL/min/1.73m2.

Any disease, concomitant injury, such as significant traumatic brain injury, or other condition that could interfere with the performance or interpretation of the protocol specified assessments, in the opinion of the investigator.

Any other social or medical condition (e.g., uncontrolled diabetes, unstable hypertension) which, in the opinion of the investigator, would make the subject unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological | 12 weeks
  MEP amplitudes (corticospinal contribution) in key target muscle groups

SECONDARY OUTCOMES:
10mWT time | 12 weeks
  Walking speed
9-HPT time | 12 weeks
  Upper extremity dexterity
Dynamometry testing (pinch grip, Chronic cohort 1; hand grip, Subacute cohort 2) | 12 weeks
  Recorded force
Graded and Redefined Assessment of Strength, Sensibility, and Prehension Test | 12 weeks
  Hand function Max Score 116 points
Lower extremity motor score (LEMS) | 12 weeks
  Lower extremity Max Score 50 points
Upper extremity motor score (UEMS) | 12 weeks
  Upper extremity Max Score 50 points
Incidences of Treatment Emergent Adverse Events (Safety and Tolerability) | 16 Weeks
  incidences of treatment emergent adverse events
Plasma Concentration of Study Drug | 12 Weeks
  initial and steady state predose and peak plasma drug concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mikol, M.D. Ph.D., Study Director — NervGen Pharma
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Connect SCI Study Website — https://www.connectscistudy.com
- See also: SCI Trials Finder Website — https://scitrialsfinder.net/trials/NCT05965700